CLINICAL TRIAL: NCT00955032
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Apathy in Parkinson's Disease.
Acronym: ReStore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0004762006
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Results first posted 2012-02-20 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2012-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Apathy; rTMS; Repetitive transcranial magnetic stimulation; Depression
MeSH Terms: conditions — Parkinson Disease; Lethargy; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-Frequency Repetitive Transcranial Magentic Stimulation (Experimental): High-Frequency repetitive transcranial magnetic stimulation patients randomized to this treatment will receive left prefrontal rTMS, each treatment will consist of 2000 stimuli (50 - 8-second trains of 40 stimuli at 5 Hz). We will administer rTMS trains every 30 seconds for 25 minutes. Stimulus intensity for the first and second trains will be 80 and 90% of Motor Evoked Potential (MEP) threshold, respectively.
  Interventions: Device: High-Frequency Repetitive Transcranial Magnetic Stimulation
- Sham Repetitive Transcranial Magentic Stimulation (Sham Comparator): Sham repetitive transcranial magnetic stimulation patients randomized to receive the sham rTMS will undergo the same procedure for identifying stimulus location used in patients receiving real rTMS. Simulated rTMS will be administered using Magstim Placebo 70 mm figure-of-8 shaped coils which produce discharge noise and vibration similar to a real 70 mm coil without stimulating the cerebral cortex. However, in addition to obvious coil discharge noise, rTMS also causes electrical stimulation of the scalp. We will simulate this experience by attaching surface electrodes underneath the sham coil and in contact with the scalp.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: High-Frequency Repetitive Transcranial Magnetic Stimulation — In patients randomized to receive left prefrontal rTMS, each treatment will consist of 2000 stimuli (50 - 8-second trains of 40 stimuli at 5 Hz). We will administer rTMS trains every 30 seconds for 25 minutes. Stimulus intensity for the first and second trains will be 80 and 90% of MEP threshold, respectively.
  Other Names: rTMS Treatment
  Arms: High-Frequency Repetitive Transcranial Magentic Stimulation
Device: Sham Repetitive Transcranial Magnetic Stimulation — Patients randomized to receive sham rTMS will undergo the same procedure for identifying stimulus location used in patients receiving real rTMS. Simulated rTMS will be administered using Magstim Placebo 70 mm figure-of-8 shaped coils which produce discharge noise and vibration similar to a real 70 mm coil without stimulating the cerebral cortex. However, in addition to obvious coil discharge noise, rTMS also causes electrical stimulation of the scalp. We will simulate this experience by attaching surface electrodes underneath the sham coil and in contact with the scalp.
  Other Names: Sham Treatment
  Arms: Sham Repetitive Transcranial Magentic Stimulation

SUMMARY:
The purpose of this research study is to attempt to treat apathy in Parkinson's disease (PD) using high-frequency repetitive transcranial magnetic stimulation (rTMS) of the brain and to investigate the patterns of brain activation that may be involved in apathy. It is hypothesized that high-frequency rTMS of the left mid-dorsolateral frontal cortex will improve apathy in PD.

DETAILED DESCRIPTION:
Apathy is a syndrome characterized by a primary lack of motivation and it manifests in three domains: behavioral (lack of effort and productivity, dependence on others for structuring daily activities), cognitive (loss of interest in new experiences, lack of concern for one's problems) and affective (flattened affect and lack of response to positive or negative events). Apathy has been consistently attributed to functional disturbance of neural systems involving mesial frontal and the anterior cingulate cortex (ACC), an area with reciprocal connections with limbic, frontal cortices and the basal ganglia.

Repetitive transcranial magnetic stimulation (rTMS) is a noninvasive tool used to manipulate activity in specific brain neural circuits through the skull and, in turn, induce short-term (milliseconds) and long-term (minutes to hours) changes in behavior. The duration of effect depends on the stimulation mode. Several studies have now demonstrated that rTMS may facilitate or modulate behavior beyond the actual stimulation. rTMS of the mid-dorsolateral frontal cortex (MDLFC) has been used to treat depression presumably because of its modulatory effect on the fronto-cingulate system (MDLFC and the ACC circuitry). Studies have shown that rTMS of the left MDLFC modulates the blood flow response in the ACC. We therefore hypothesize that high-frequency rTMS of the left MDLFC will also improve apathy in PD.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of "probable" PD, defined by the presence of at least 2 out of 3 cardinal motor features of PD (resting tremor, rigidity, and bradykinesia, plus a sustained and significant response to dopaminergic treatment);
2. age 30 or over; and
3. on stable medications for at least 30 days.

Exclusion Criteria:

1. features suggestive of other causes of parkinsonism/ parkinson-plus syndromes;
2. history of deep brain stimulation or ablation surgery, significant headaches, epilepsy or seizure disorder, mass brain lesions, or major head trauma leading to loss of consciousness of any length;
3. family (1st degree relatives) history of epilepsy;
4. evidence for dementia;
5. presence of contraindications for functional magnetic resonance imaging (fMRI);
6. history of schizophrenia, schizoaffective disorder, other psychosis, rapid-cycling bipolar illness, alcohol/drug abuse within the past year;
7. need for rapid clinical response due to conditions such as initiation, psychosis, or suicidality;
8. unstable medical condition such as diabetes, cardiac disease, hypertension;
9. pregnancy; and
10. colorblindness.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hubert H Fernandez, M.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- See also: Movement Disorders Center at the University of Florida — http://mdc.mbi.ufl.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients seen clinically for routine clinical care were determined by clinicians if they appeared to qualify for the study. Subjects were asked and consented in a non-coercive manner if they wished to be contacted via telephone about future study participation. Recruitment occurred between March 2007-December 2009.
Groups:
- rTMS Treatment: Participants in this group received rTMS treatment.
- Sham Treatment: Participants in this group did not receive rTMS treatment.
Period: Overall Study
Arm/Group | rTMS Treatment | Sham Treatment
Started | 16 | 8
Completed | 16 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rTMS Treatment | Sham Treatment | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 0 | 10
  >=65 years | 6 | 8 | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 63.8 (7.2) | 72.8 (5.7) | 66.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 14 | 5 | 19
Region of Enrollment [Number; unit: participants]
  United States | 16 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Apathy Evaluation Scale (AES)
Description: The apathy evaluation scale is a 14-item self-report questionaire that provides a quantitative estimate of apathy symptoms. Items are given a score of 0-3, and a total score is summated using all items. Scores may range between 0 and 42. Higher scores are indicative of greater symptoms of apathy, and a score of 14 is suggestive of clinically significant symptoms.
Time Frame: Pre-Tx; 10 days post tx
Population: All participants who completed study procedures were included for analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- rTMS Pre TX: Participants in this group were assessed prior to rTMS treatment.
- Sham Pre TX: Participants in this group were assessed before sham treatment.
- rTMS Post TX (Immediate): Participants in this group received rTMS treatment and were assessed approximately 10 days after tx began.
- Sham Post Tx (Immediate): Participants in this group did not receive rTMS treatment and were assessed approximately 10 days after tx began.
Arm/Group | rTMS Pre TX | Sham Pre TX | rTMS Post TX (Immediate) | Sham Post Tx (Immediate)
Number analyzed (Participants) | 16 | 8 | 16 | 8
units on a scale | 19.6 (5.1) | 18.8 (3.9) | 17.9 (7.0) | 16.8 (4.6)

2. Secondary Outcome: Lille Apathy Rating Scale (LARS)
Description: The Lille Apathy Rating Scale (LARS) is a 33-item interviewer administered structured questionaire designed to assess level of apathetic symptoms. The first 3 items are scored from -2 to +2, while the remainder items are scored from -1 to +1. Scores can range between -36 to +36. The more positive the score, the greater level of apathy symptoms.
Time Frame: Pre-Tx; 10 days post-tx
Population: All participants who completed study procedures were included for analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- rTMS Pre tx: Participants in this group received were assessed prior to receiving rTMS treatment.
- Sham Pre tx: Participants in this group were assessed prior to receiving Sham treatment.
- rTMS Post tx: Participants in this group received rTMS treatment and were assessed approximately 10 days after tx began.
- Sham Post tx: Participants in this group did not receive rTMS treatment and were assessed approximately 10 days after tx began.
Arm/Group | rTMS Pre tx | Sham Pre tx | rTMS Post tx | Sham Post tx
Number analyzed (Participants) | 16 | 8 | 16 | 8
units on a scale | -15.6 (9.1) | -18.9 (4.5) | -20.1 (7.8) | -22.1 (5.2)

3. Secondary Outcome: Beck Depression Inventory-Second Edition (BDI-II)
Description: The Beck Depression Inventory-Second Edition (BDI-II) is a 21-item self-report questionaire that measures depressive symptoms. Each item is scored on a scale of 0-3, and items are summated to yield a total score. A higher score is indicative of greater symptoms of depression. Total scores may range between 0 and 63. A score greater than or equal of 14 is suggestive of clinically significant symptoms.
Time Frame: Pre-Tx; 10 days post-tx
Population: All participants who completed study procedures were included for analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- rTMS Pre tx: Participants in this group were assessed before they received rTMS treatment.
- Sham Pre tx: Participants in this group were assessed before they received Sham tx.
Arm/Group | rTMS Pre tx | Sham Pre tx | rTMS Post tx | Sham Post tx
Number analyzed (Participants) | 16 | 8 | 16 | 8
units on a scale | 17.1 (8.4) | 17.8 (9.8) | 11.8 (8.8) | 11.8 (5.4)

4. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D)
Description: The Hamilton Depression Rating Scale (HAM-D) is a 24-item interviewer administered structure questionaire designed to assess symptoms of depression. Items are scored with a range of 0-4, though 11 of the items are scored between 0 and 2. A total score is then calculated of all items which can range from 0 to 74. A higher score is indicative of more depressive symptoms, and a lower score post-tx is indicative of better outcome.
Time Frame: Pre-Tx; 10 days post-tx
Population: All participants who completed study procedures were included for analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sham Pre tx: Participants in this group were assessed before they received sham treatment.
Arm/Group | rTMS Pre tx | Sham Pre tx | rTMS Post tx | Sham Post tx
Number analyzed (Participants) | 16 | 8 | 16 | 8
units on a scale | 12.5 (7.3) | 11.9 (6.5) | 7.9 (4.8) | 8.5 (5.4)

ADVERSE EVENTS:
Time Frame: Adverse event data were collect from study enrollment to study completion, which occured between March 2007 - December 2009.
Arm/Group | rTMS Treatment | Sham Treatment
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/8
Other Adverse Events (participants affected / at risk) | 8/16 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rTMS Treatment (N=16) | Sham Treatment (N=8)
Falling (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rTMS Treatment (N=16) | Sham Treatment (N=8)
Headache (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Hallucination (General disorders) | 0 (0) | 1 (1)
Back Pain (General disorders) | 1 (1) | 1 (1)
Worsening PD symptoms (General disorders) | 3 (3) | 0 (0)
Fall (General disorders) | 2 (2) | 0 (0)
Pitting Edema (General disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to recruiting difficulties, only 24 participants completed study participation. Despite this, the investigators still had significant power to examine effects of interest.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No